CLINICAL TRIAL: NCT01375387
Title: A Phase I, Randomized Double-blind, Placebo-controlled, Single-center, Single-dose, Three-way Cross-over Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Lacosamide Tablets in Healthy Male Chinese and Japanese Subjects
Brief Title: Three-way-cross-over Study to Evaluate Safety and Pharmacokinetics of Lacosamide in Healthy Japanese and Chinese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SP1046; 2010-023164-40 (EudraCT Number)
Record Dates: First submitted 2011-04-19; First posted 2011-06-17 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers
Keywords: Vimpat; Pharmacokinetics; Healthy Japanese male; Healthy Chinese male
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Lacosamide 100 mg, Japanese (Experimental): 1 Lacosamide 100 mg tablet plus 3 placebo tablets
  Interventions: Drug: Lacosamide; Other: Placebo 3
- Lacosamide 100 mg, Chinese (Experimental): 1 Lacosamide 100 mg tablet plus 3 placebo tablets
  Interventions: Drug: Lacosamide; Other: Placebo 3
- Lacosamide 200 mg, Japanese (Experimental): 2 Lacosamide 100 mg tablets plus 2 placebo tablets
  Interventions: Drug: Lacosamide; Other: Placebo 2
- Lacosamide 200 mg, Chinese (Experimental): 2 Lacosamide 100 mg tablets plus 2 placebo tablets
  Interventions: Drug: Lacosamide; Other: Placebo 2
- Lacosamide 400 mg, Japanese (Experimental): 4 Lacosamide 100 mg tablets
  Interventions: Drug: Lacosamide
- Lacosamide 400 mg, Chinese (Experimental): 4 Lacosamide 100 mg tablets
  Interventions: Drug: Lacosamide
- Placebo Comparator, Japanese (Placebo Comparator): 4 placebo tablets
  Interventions: Other: Placebo 4
- Placebo Comparator, Chinese (Placebo Comparator): 4 placebo tablets
  Interventions: Other: Placebo 4

INTERVENTIONS:
Drug: Lacosamide — 100 mg oral tablet, single dose
  Other Names: Vimpat®
  Arms: Lacosamide 100 mg, Chinese; Lacosamide 100 mg, Japanese
Drug: Lacosamide — Lacosamide 2 X 100 mg tablet
  Other Names: Vimpat®
  Arms: Lacosamide 200 mg, Chinese; Lacosamide 200 mg, Japanese
Drug: Lacosamide — Lacosamide 4 X 100mg tablet
  Other Names: Vimpat®
  Arms: Lacosamide 400 mg, Chinese; Lacosamide 400 mg, Japanese
Other: Placebo 3 — Placebo - 3 tablets
  Arms: Lacosamide 100 mg, Chinese; Lacosamide 100 mg, Japanese
Other: Placebo 4 — Placebo - 4 tablets
  Arms: Placebo Comparator, Chinese; Placebo Comparator, Japanese
Other: Placebo 2 — Placebo - 2 tablets
  Arms: Lacosamide 200 mg, Chinese; Lacosamide 200 mg, Japanese

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of lacosamide following single oral administration of lacosamide 100 mg, 200 mg and 400 mg in healthy male Chinese and Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese or Japanese volunteers

Exclusion Criteria:

* Subject has participated or is participating in any other clinical studies of Lacosamide within the last 3 months
* Subject is not healthy (eg, taking any drug treatments, excessive amount of alcohol, cigarettes or caffeine, having any psychological or emotional problems, a drug/alcohol abuse, abnormal diet, having abnormal safety parameters)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) of lacosamide in plasma. | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Area under the curve from 0 to the time of the last quantifiable concentration (AUC(0-t)) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Area under the curve from 0 to infinity (AUC) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (tmax) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Terminal half-life (t½) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Apparent total body clearance (CL/F) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Apparent volume of distribution (Vz/F) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Mean resident time (MRT) of lacosamide in plasma. | Multiple sampling from 0 to 72 hours following single dose in each treatment period
First order terminal elimination rate constant (λZ ) of lacosamide in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Maximum drug concentration (Cmax) of SPM12809 in plasma. | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Area under the curve from 0 to the time of the last quantifiable concentration (AUC(0-t)) of SPM12809 in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Area under the curve from 0 to infinity (AUC) of SPM12809 in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Time to reach maximum plasma concentration (tmax) of SPM12809 in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Terminal half-life (t½) of SPM12809 in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
First order terminal elimination rate constant (λZ ) of SPM12809 in plasma | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Total amount of drug excreted in urine (Ae) of lacosamide and SPM12809 | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Fraction of dose excreted in urine (fe) of lacosamide and SPM12809 | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Renal clearance (CLR) of lacosamide and SPM12809 | Multiple sampling from 0 to 72 hours following single dose in each treatment period
Apparent formation clearance of metabolites (CLfm/F) | Multiple sampling from 0 to 72 hours following single dose in each treatment period
AUC Ratio | Multiple sampling from 0 to 72 hours following single dose in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Neuss, Germany